CLINICAL TRIAL: NCT00911014
Title: Access to Healthcare, Patient Comprehension and Future Plans of Women Undergoing Surgery for a Vesicovaginal Fistula in Niamey, Niger
Status: Completed | Type: Observational
Sponsor: Ascher-Walsh, Charles, M.D. (Individual)
Responsible Party: Charles Ascher-Walsh, MD, Mount Sinai School of Medicine
Other Study IDs: HSD08-00564
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Vesicovaginal Fistula; Delivery of Healthcare
MeSH Terms: conditions — Vesicovaginal Fistula | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vesicovaginal fistula repair: Women undergoing repair of vesicovaginal fistula
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — From September 2005 to January 2006, 58 women who underwent surgery for vesicovaginal fistula at the National Hospital Fistula Center in Niamey, Niger were interviewed post-operatively using a questionnaire developed to investigate demographic, social, economic, and cultural factors that may affect formation of fistula. Also included in this questionnaire was evaluation of access to health care as well as patient understanding of counseling regarding their surgery and post-operative instructions, in particular information about future fertility and fistula development.

SUMMARY:
Evaluate access to healthcare, comprehension of pre-operative counseling and post-operative goals of women treated for vesicovaginal fistula in Niger through use of a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent surgery for repair or vesicovaginal fistula

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women who underwent surgery for repair of vesciovaginal fistula in Niamey, Niger
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2005-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Access to healthcare | 1 year

SECONDARY OUTCOMES:
Comprehension of pre-operative counselling | 1 year
Post-operative goals of women undergoing repair of vesicovaginal fistula | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ascher-Walsh, MD, MS, Study Director — Mt Sinai School of Medicine, Dept Obstetrics and Gynecology
Locations (1):
- Mount SInai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Meyer L, Ascher-Walsh CJ, Norman R, Idrissa A, Herbert H, Kimso O, Wilkinson J. Commonalities among women who experienced vesicovaginal fistulae as a result of obstetric trauma in Niger: results from a survey given at the National Hospital Fistula Center, Niamey, Niger. Am J Obstet Gynecol. 2007 Jul;197(1):90.e1-4. doi: 10.1016/j.ajog.2007.03.071. PMID 17618772